CLINICAL TRIAL: NCT05970822
Title: A Phase 1b Study Evaluating Safety, Pharmacokinetics, Pharmacodynamics and Efficacy of BC3402 in Combination With Azacitidine in Subjects With Myelodysplastic Syndrome (MDS) and Chronic Myelomonocytic Leukemia (CMML)
Brief Title: Study of BC3402 in Combination With Azacitidine in Patients With MDS and CMML
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Biocity Biopharmaceutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BC3402-104
Record Dates: First submitted 2023-07-13; First posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Myelodysplastic Syndromes; Chronic Myelomonocytic Leukemia
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic | interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BC3402+azacitidine (Experimental): Subjects will receive azacitidine and BC3402 in a treatment cycle.
  Interventions: Drug: BC3402; Drug: Azacitidine

INTERVENTIONS:
Drug: BC3402 — Escalating of BC3402 will be administered IV(intravenous)
Drug: Azacitidine — Azacitidine will be administered daily

SUMMARY:
The study is to evaluate safety, pharmacokinetics, pharmacodynamics and efficacy of BC3402 in combination with azacitidine (AZA) in subjects with Myelodysplastic Syndrome (MDS) and Chronic myelomonocytic leukemia (CMML)

ELIGIBILITY:
Inclusion Criteria:

1. MDS and CMML subjects with higher risk;
2. Age ≥ 18 years old;
3. Eastern Cooperative Oncology Group score of 0~2;
4. Not suitable for or refuse to receive hematopoietic stem cell transplant(HSCT);
5. Subjects should take effective contraceptive measures
6. Must sign the Informed Consent Form (ICF), and be able to follow all study procedures.

Exclusion Criteria:

1. Prior exposure to anti-TIM-3 therapy at any time
2. Previous HSCT
3. Live vaccine administered within 4 weeks prior to start of treatment
4. Current use or use within 7 days prior to start of treatment of systemic steroid therapy (> 10 mg/day prednisone or equivalent) or any immunosuppressive therapy. Topical, inhaled, nasal, ophthalmic steroids are allowed.

Other protocol-defined Inclusion/Exclusion may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-06-18 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with AEs and SAEs Primary endpoint:Incidence of dose limiting toxiecities(DLTs) and incidence of DLT events within 28 days (first cycle) | 2.5 years
  To evaluate the safety and tolerability of BC3402

CONTACTS AND LOCATIONS:
Overall Officials: Zhijian Xiao, MD, Principal Investigator — Chinese Academy of Medical Sciences
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality, China